CLINICAL TRIAL: NCT01677845
Title: Phase I Study of Hypo-Fractionated Radiation Therapy (HRT) for Localized Prostate Cancer
Brief Title: Hypo-Fractionated Radiation Therapy for Localized Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI no longer with the institution
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-00867
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: Localized Prostate Cancer; Radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy (Experimental): Radiation Therapy
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Dose Level 1: 54 Gy; 3 Gy per fraction; 3 days per week x 6 weeks for a total of 18 fractions;
  Dose Level 2: 55.8 Gy; 3.1 Gy per fraction; 3 days per week x 6 weeks for a total of 18 fractions;
  Dose Level 3: 57.6 Gy; 3.2 Gy per fraction; 3 days per week x 6 weeks for a total of 18 fractions.

SUMMARY:
The aim of this study is to determine the maximum tolerated dose of hypo-fractionated radiation therapy and the toxicity of the treatment program.

Eligible patients with stage T1-2c prostate cancer who sign consent will be enrolled to this phase I dose escalation trial and be treated with hypo-fractionated radiation therapy (HRT). Dose escalation will be as follows:

There will be 3 cohorts consisting of 3 patients each.

DETAILED DESCRIPTION:
Dose escalation will be as follows:

There will be 3 cohorts consisting of 3 patients each. All patients will receive 18 fractions of HRT over the course of 6 weeks (3 fractions per week). Dose level I will be 54Gy (3 Gy per fraction), dose level II will be 55.8 Gy (3.1Gy per fraction), dose level III will be 57.6 Gy (3.2 Gy per fraction). After accrual of dose level I, all patients will be observed for a minimum of two weeks after completion of radiation treatments, for assessment of toxicity, before the dose can be escalated for the next cohort. After dose level II, patients will be observed for 6 months before enrolling patients on dose level III.

All patients will be seen weekly by their radiation oncologist during radiation therapy. Any observations regarding radiation reactions will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* History/physical examination with digital rectal examination of the prostate within 8 weeks prior to registration
* Clinical stage T1-2c (AJCC 6th edition)
* Gleason <6 and PSA <10 ng/mL
* Gleason =7 and/or PSA 10-20 ng/mL provided <34% of core biopsies are positive for carcinoma
* PSA < 20 ng/mL within 180 days prior to registration. PSA should not be obtained for at least 10 days after prostate biopsy.
* Zubrod performance status 0-1
* Age ≥ 18
* Patient must sign study specific informed consent prior to randomization.

Exclusion Criteria:

* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years. (For example, carcinoma in situ of the bladder or oral cavity is permissible)
* Evidence of distant metastases
* Regional lymph node involvement
* Previous radical surgery (prostatectomy) or cryosurgery for prostate cancer
* Prior androgen deprivation therapy (ADT)
* Previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* Previous or concurrent cytotoxic chemotherapy for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-05; Primary Completion 2017-02 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
the maximum tolerated dose of HRT | 30 weeks
  After accrual of dose level I, all patients will be observed for a minimum of two weeks after completion of radiation treatments, for assessment of toxicity, before the dose can be escalated for the next cohort. After dose level II, patients will be observed for 6 months before enrolling patients on dose level III.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Sanfilippo, MD, Principal Investigator — NYU Langone Medical Center, Departement of Radiation Oncology
Locations (1):
- NYU Langone Medical Center, New York, New York, United States